CLINICAL TRIAL: NCT01560793
Title: Phase I Study of the Safety and Immunogenicity of a Novel H5N1 Influenza Vaccine in Healthy Adults Age 18-49 Years
Brief Title: Safety and Immunogenicity of a Novel H5N1 Influenza Vaccine in Healthy Adults Age 18-49 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: VAX161-01B
Record Dates: First submitted 2012-02-14; First posted 2012-03-22 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: Influenza; Vaccines; H5N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VAX161B (Experimental): Dose escalating study where subjects are treated with VAX161B at one of six dose levels. Subjects will be injected with VAX161B twice during the study at Day 0 and Day 21. The dosages are: 1 mcg; 2.5 mcg; 4 mcg; 6 mcg; 8 mcg; and 12 mcg.
  Interventions: Biological: VAX161 [STF2.HA5 H5N1]

INTERVENTIONS:
Biological: VAX161 [STF2.HA5 H5N1] — dose escalating, 2 intramuscular doses given 21 days apart

SUMMARY:
This study will evaluate the safety and immunogenicity of VAX161B [STF2.HA5 H5N1], a recombinant, inactivated, subunit influenza vaccine given as a two dose regimen at a range of doses.

DETAILED DESCRIPTION:
The purpose of this study is to test an investigational vaccine known as "VAX161B". VAX161B is a vaccine for the influenza A virus subtype H5N1 avian influenza virus (bird flu). In this study, the subject will receive the VAX161B vaccine at one of five doses to see which does might be the best. VaxInnate want to find out how safe these vaccines are and how well they are tolerated by people who receive them. To measure how effective each type of vaccine is, VaxInnate will test the ability of the body to develop an immune response, which means how well the body recognizes and defends itself against the influenza virus.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18 - 49 years inclusive
* give written informed consent to participate
* healthy, as determined by medical history, physical examination
* comprehension of the study requirements
* willing to provide multiple blood specimens collected by venipuncture.

Exclusion Criteria:

* Subjects who have a psychiatric illness, a chronic illness that would interfere with participation or interpretation of results
* clinically significant abnormal liver function tests
* positive serology for HBsAg or HCV antibodies
* impaired immune responses
* history of anaphylactic type reaction to injected vaccines
* history of drug or chemical abuse in the year prior to screening
* history of Guillain-Barré Syndrome
* history of chronic obstructive pulmonary disease or history of other lung disease

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  Assess safety, reactogenicity and tolerability. Symptoms will be collected from the memory aid and from the information collected at the clinic visits. All symptoms will be graded according to severity. Response to vaccine will be categorized as local (arm pain, redness, bruising, etc.) or systemic (headache, muscle aches, fatigue, etc.) symptoms. Laboratory tests such as CRP, WBC, LFTs and cytokines collected before and after vaccination will also be analyzed. We will compare the types and severity of symptoms and laboratory results based on vaccine dose.

SECONDARY OUTCOMES:
Immunogenicity | 6 mos.
  To assess serum immune response, sera collected at Days 0, 21, 42 and 180 will be analyzed for HAI, MN, serum IgG anti-HA and serum IgG anti-flagellin by Elisa. The geometric mean, seroconversion and seroprotection rates will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associates; Casey Johnson, DO, Principal Investigator — Johnson County Clin-Trials
Locations (2):
- United States (2):
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas